CLINICAL TRIAL: NCT03978702
Title: Pancreatic Surgery: Evaluation of the Impact of Pancreatectomy on Systemic Immunity
Brief Title: Evaluation of the Impact of Pancreatectomy on Systemic Immunity
Acronym: IMMUNOPANC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IMMUNOPANC-IPC 2018-051
Record Dates: First submitted 2019-06-03; First posted 2019-06-07 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-05

CONDITIONS: Pancreas Cancer; Pancreatectomy; Hyperglycemia
Keywords: Pancreatectomy; Immune system
MeSH Terms: conditions — Pancreatic Neoplasms; Hyperglycemia | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Indication for pancreatectomy (Experimental): Blood sampling at different time points before and after pancreatectomy
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — 20 mL will be collected at each time point (day-1,day 0, day 1, day 3, day 7, 1 year after pancreatectomy)

SUMMARY:
The study aims at establishing the profile of the immune reaction that occurs in the early surgical suites after pancreatectomy. Blood samples will be collected before surgery, (Day-1), at day0, and after surgery at Day 1, Day 3, Day 7 at 1 year after pancreatectomy. Mass cytometry, genomic and transcriptomic approaches will be used to evaluate the immune systemic modulation after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient with an indication of pancreatectomy
* Signed consent form

Exclusion Criteria:

* Neoadjuvant treatment
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2022-07-27 (Estimated); Study Completion 2022-07-27 (Estimated)

PRIMARY OUTCOMES:
Measurement of immune effectors (Tcells, NK) levels after pancreatectomy | 1 year
  Evaluation of immune effectors my mass cytometry after pancreatectomy (compared to baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Turrini, MD ¨PhD, Principal Investigator — Institut Paoli-Calmettes
Locations (1):
- Institut Paoli Calmettes, Marseille, France